CLINICAL TRIAL: NCT01571765
Title: Scaling Up Maternal and Child Health In Bushenyi and Rubirizi Districts, UGANDA
Brief Title: MNCH Programming in Southwest Uganda Maternal and Child Health In Bushenyi and Rubirizi Districts, UGANDA
Acronym: HCUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian International Development Agency (Other Government)
Responsible Party: Principal Investigator, Jennifer L. Brenner, Clinical Associate Professor, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIDA S-065346
Record Dates: First submitted 2012-03-30; First posted 2012-04-05 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Child Mortality; Maternal Mortality (All Cause)
Keywords: maternal; newborn; child
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MNCH programming (Experimental): protocols and training for data collection, referrals, and management for health district. Training in obstetrics, newborn care and management of sick children for health workers, Increased community health promotion such as training of CHWs, health centre management teams and bednet distribution
  Interventions: Other: MNCH programming in health district
- no added MNCH activities (No Intervention)

INTERVENTIONS:
Other: MNCH programming in health district — training at health district level in management, data collection. Training at health centres in obstetrics and pediatrics and training in community of CHWs and bednet distribution
  Arms: MNCH programming

SUMMARY:
The investigators will assess whether in Bushenyi District in southwestern Uganda, a two year intervention providing comprehensive MNCH programming will:

* Reduce morbidity and mortality for children under five years old and;
* Improve access to maternal health services Compared to a control community without MNCH intervention?

Hypothesis:

Comprehensive maternal, newborn and child health programming in Bushenyi Distrcit can have a positive impact on morbidity and mortality for children under five years and will improve access for women to maternal health services which may lead, in the longer term, to decreased maternal mortality.

DETAILED DESCRIPTION:
A detailed impact assessment will be carried out for the duration of the MNCH training and support initiative in Bushenyi District, using mixed methods. The study will assess 8 of the 11 key core MNCH indicators as identified by CIDA as a priority. Other information to be collected such as demographics and patterns of health care use, and prevalence of disease will help health planners in the districts, and will be helpful in sub analysis and interpretation of findings. The main study will use household surveys in both districts at baseline, midline and endline. Other tools will include pre and post qualitative surveys (FGDs, KII) and analysis of operational data.

The main study group will be representative communities and health centres within Bushenyi District who will receive intervention between 2012 and 2014; Rubirizi District will serve as a control area for this study but will received selected MNCH services starting in 2013 after midline data are collected.

ELIGIBILITY:
Inclusion Criteria:

* all households living in selected communities; all women 15-49 living in selected communities Exclusion Criteria: none

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10985 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Reduced morbidity for children under five years old | 2 years

SECONDARY OUTCOMES:
improved maternal access to health services | 24 months
  proportion of pregnant women who have attended antenatal care four or more times; proportion of women whose most recent delivery was attended by a skilled birth attendant; met need for contraception (CIDA indicator)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brenner, MD, Principal Investigator — University of Calgary; Jerome Kabakyenga, MBBS, PHD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Mbarara, Uganda